CLINICAL TRIAL: NCT02355249
Title: Traditional Three Incisions vs Minimally Invasive Thoracol-laparoscopic Esophagectomy for Esophageal Cancer: a Multi-center, Randomized, and Open-label Trial
Brief Title: Traditional Three Incisions vs Minimally Invasive Thoracol-laparoscopic Esophagectomy for Esophageal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: China-Japan Friendship Hospital (Other); Peking University Cancer Hospital & Institute (Other); Beijing Chao Yang Hospital (Other); Peking University Third Hospital (Other); The Second People's Hospital of Sichuan (Other); First Affiliated Hospital of Chongqing Medical University (Other); Hunan Cancer Hospital (Other); The Affiliated Tumor Hospital of Nantong University, Nantong, Jiangsu Province, China (Other); First Hospital of China Medical University (Other); Quanzhou First Hospital (Other); Jiangxi Provincial People's Hopital (Other); People's Hospital of Guangxi Zhuang Autonomous Region (Other)
Responsible Party: Principal Investigator, Jie He, M.D. & Ph.D. , President of CICAMS, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201412
Record Dates: First submitted 2015-01-26; First posted 2015-02-04 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-01

CONDITIONS: Esophageal Carcinoma
Keywords: traditional three incisions; minimally invasive thoracol-laparoscopic esophagectomy; MIE; esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A group (MIE) (Experimental): Via minimally invasive thoracol-laparoscopic esophagectomy.
  Interventions: Procedure: MIE
- B group (OE) (Active Comparator): Via traditional three incisions esophagectomy.
  Interventions: Procedure: OE

INTERVENTIONS:
Procedure: MIE — Minimally invasive thoracol-laparoscopic esophagectomy will be performed in this group.
  Arms: A group (MIE)
Procedure: OE — Patients will be treated with traditional three incisions esophagectomy.
  Arms: B group (OE)

SUMMARY:
This study is a multi-center, randomized, and open-label trial to compare the safety and feasibility of traditional three incisions and minimally invasive thoracol-laparoscopic esophagectomy for esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of intrathoracic esophageal carcinoma of Stage I to III, which is potentially resectable judged by MDT
2. 18≤age≤75
3. cT1b-4a，N0-2，M0 confirmed by chest CT, EUS, or EUS-FNA in four weeks;
4. ECOG PS scores≤2
5. Laboratory findings in 14 days before operation：normal blood test of basic metabolism panel
6. European Clinical Oncology Group (ECOG) performance status 0,1 or 2
7. More than 12 months of expected survival
8. Tolerance of tracheal intubation and general anesthesia
9. Written informed consent

Exclusion Criteria:

1. Carcinoma of the cervical esophagus or gastro-esophageal junction (GEJ)
2. Prior thoracic surgery which may effect this study
3. Pregnant or breast feeding
4. Inability to tolerance of tracheal intubation and general anesthesia
5. PS >2
6. unstable disease
7. Poor compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 648 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of respiratory complications | 1 months
  Respiratory complications including respiratory failure requiring mechanical ventilation, atelectasis needs suctioning of bronchoscopy, lung infection needs medication, adult respiratory distress syndrome.

SECONDARY OUTCOMES:
Short-term Effects of Traditional Three Incisions Surgery vs Minimally Invasive Thoracol-laparoscopic Esophagectomy for Esophageal Cancer | 2 years
  To observe differences of short-term effects(bleeding volume during operation,operation time, hospital mortality, 2 years DFS) between two groups.
The incidence of postoperative complications except respiratory complications | 1 months
  Surgical Complications except respiratory complications(such as infection, esophageal fistula, etc.) will be measured by the Clavien-Dindo Classification
lung function | before operation, 1, 3 months after surgery
  lung function will be measured by VC,FVC,FEV1,DLCO
Pain Scores after surgery | before operation, 1, 3 days and 1, 3, 6 months after surgery
  Pain Scores will be measured by Brief pain inventory(BPI)
Health-related quality of life scores（HRQoL） | before operation, 1, 3, 6, 9, 12, 15,18, 21, 24 months after surgery
  HRQoL will be measured by EORTC QLO-C30, QLQ-OES18

OTHER OUTCOMES:
blood biomarker analysis | 1 months
  The presence of inflammatory factors and stress response indicators (ATCH, C- reactive protein, interleukin-6, etc.)of esophageal tissue specimens and blood samples will be explored

CONTACTS AND LOCATIONS:
Overall Officials: Jie He, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (13):
- China (13):
  - Cancer Hospital of Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - China-japan friendship hospital, Beijing, Beijing Municipality
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Chao-Yang Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Quanzhou First Hospital, Quanzhou, Fujian
  - The People's Hospital Of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The Second People's Hospital of Sichuan, Chengdu, Sichuan

REFERENCES:
- [Derived] Mu J, Gao S, Mao Y, Xue Q, Yuan Z, Li N, Su K, Yang K, Lv F, Qiu B, Liu D, Chen K, Li H, Yan T, Han Y, Du M, Xu R, Wen Z, Wang W, Shi M, Xu Q, Xu S, He J. Open three-stage transthoracic oesophagectomy versus minimally invasive thoraco-laparoscopic oesophagectomy for oesophageal cancer: protocol for a multicentre prospective, open and parallel, randomised controlled trial. BMJ Open. 2015 Nov 17;5(11):e008328. doi: 10.1136/bmjopen-2015-008328. PMID 26576807